CLINICAL TRIAL: NCT04324892
Title: Effects of Achieving SDAI Remission on Joint Space Outcomes Progression in Early Rheumatoid Arthritis: an HR-pQCT Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.224
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Treat to target; HRpqCT; Joint space narrowing; SDAI remission
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treat to target: The study has only 1 cohort with treat-to-target strategy
  Interventions: Drug: Treat to target

INTERVENTIONS:
Drug: Treat to target — All patient will received protocolized treatment with an aim to achieve SDAI remission

SUMMARY:
Objectives:

To elucidate the effects of achieving sustained simple disease activity index (SDAI) remission in the progression of joint space outcomes using high-resolution peripheral quantitative CT (HR-pQCT) in patients with early rheumatoid arthritis (ERA), and what the independent effects of erosion /JSW progression are on patient's function.

Hypothesis to be tested: Effective control of inflammation in ERA patients who can achieve sustained SDAI remission will have less progression of joint damage then patients who cannot achieve sustained SDAI remission.

Design and subjects: 110 consecutive ERA patients will participate in this 1-year prospective, hospital-based, cohort study.

Study instruments Metacarpophalangeal joints 2-4 will be measured using HR-pQCT Interventions All participants will receive 1-year tight-control treatment according to a standardized protocol aiming at SDAI remission. Physical function will be assessed by Health Assessment Questionnaire (HAQ) at each visit. HR-pQCT and radiographs will be performed at baseline, 6 (HR-pQCT only) and 12 months. Quantitative analysis of joint space width (JSW) and volume, erosion number and volume, and marginal osteosclerosis (bone apposition at the base of the erosion) will be evaluated by HR-pQCT. Radiographic progression will be scored using van der Heijde-Sharp (SvdH) score.

Outcome measures: The primary outcome is the change in JSW and volume over a period of 12 months. Main secondary outcomes include changes in the i) number and size of erosion, ii) SvdH score and iii) HAQ over a period of 12 months.

Expected results: Patients who can achieve sustained SDAI remission will have less joint damage and functional loss compared

ELIGIBILITY:
Inclusion Criteria:

* fulfilled the 2010 ACR/EULAR classification criteria for RA
* have symptoms onset of less than 2 years,
* have active disease (SDAI >3.3)

Exclusion Criteria:

* have severe clinical deformity at the 2nd, 3rd or 4th MCP joint which precluded a reliable HR-pQCT examination and resulted in motion artefacts influencing the scanning accuracy
* are pregnant or breast feeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Starting from July 2020, all new cases referrals to the rheumatology clinic of the Prince of Wales Hospital (PWH) and four other regional hospitals in Hong Kong will be screened by a research assistant. Patients referred as RA, possible RA or undifferentiated arthritis will be contacted through telephone. Patients with at least 1 tender and swollen joint and with duration of symptoms less than 2 years and with no previous use of DMARDs will be invited to a screening visit at the early arthritis clinic of the PWH within 2 weeks of the referral, where they will be formally assessed by a rheumatologist.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-07-12 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Effect of achieving Sustained SDAI remission (SDI group) on the progression of joint space size and volume compared to those who cannot achieve sustained SDAI remission (non-SDI group) | 12 months
  To study the effect of achieving Sustained SDAI remission at 6, 9 and 12 months (SDI group) on the progression of joint space size and volume over a period of 12 months as evaluated by HR-pQCT compared to those who cannot achieve sustained SDAI remission (non-SDI group)

SECONDARY OUTCOMES:
Changes in size of erosion and marginal osteosclerosis using HR-pQCT, and SvDH score at 12 months between the SDI group and non-SDI group | 12 months
  To study the changes in size of erosion and marginal osteosclerosis using HR-pQCT, and SvDH score by convention X-ray at 12 months between the SDI group and non-SDI group
Changes in joint space and erosion size as a function of inflammatory activity as reflected by the time-averaged SDAI. | 12 months
  To investigate the changes in joint space and erosion size as a function of inflammatory activity as reflected by the time-averaged SDAI.
Association between the changes in joint space and erosion size on HR-pQCT and HAQ-DI | 6 months
  To investiage the association between the changes in joint space and erosion size on HR-pQCT and HAQ-DI to determine the impact of joint damage on reversible and non-reversible disability.
Association between the changes in joint space and erosion size on HR-pQCT and HAQ-DI | 12 months
  To investiage the association between the changes in joint space and erosion size on HR-pQCT and HAQ-DI to determine the impact of joint damage on reversible and non-reversible disability.
Association between the changes in SvdH score and HAQ-DI over a period 12 months | 12 months
  To investigate the association between the changes in SvdH score and HAQ-DI

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hopsital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No